### **Informed Consent Form**

Version/Approval Date (Güncelleme/Onay Tarihi): 01/07/2024

#### PLEASE TAKE TIME TO READ THIS DOCUMENT CAREFULLY

You are invited to participate in the study titled "Evaluation of the Effectiveness of a Web-Based Breastfeeding Education Program Based on the Information-Motivation-Behavioral Skills (IMB) Model", conducted by Ömür Aktaş under the supervision of Prof. Dr. Sena Kaplan.

Before deciding whether to participate, it is important that you understand **why and how the study will be conducted**. Therefore, reading and understanding this form is crucial. If you do not understand any part of this form or would like more information, please ask the research team.

Participation in this study is entirely **voluntary**. You have the right **not to participate**, or to **withdraw from the study at any time**. Completing the study materials will be interpreted as giving your consent to participate. You should answer the questions freely without any pressure or influence. The information obtained from these forms will be used **solely for research purposes**.

## 1. Study Information

### a. Purpose of the Study:

This study is planned as a **Randomized Controlled Experimental Study** to evaluate the effectiveness of a web-based breastfeeding education program based on the **Information-Motivation-Behavioral Skills (IMB) Model**. The study aims to examine the effect of this program on **breastfeeding self-efficacy, motivation, breastfeeding problems, and exclusive breastfeeding** in primiparous women.

## b. Study Content:

Data will be collected using the following tools:

- Individual Information Form
- Breastfeeding Knowledge Test
- Antenatal Breastfeeding Self-Efficacy Scale
- Postnatal Breastfeeding Self-Efficacy Scale
- Visual Analog Scale (VAS Motivation)
- Breastfeeding Motivation Scale
- Breastfeeding Problems Assessment Scale

- Postpartum Follow-Up Form-1 and Postpartum Follow-Up Form-2
- c. Reason for the Study:
  - Scientific Research
  - Thesis Study
- d. Estimated Duration: Approximately 30 minutes
- e. Expected Number of Participants/Volunteers: 70
- **f. Study Location(s):** Gazi University Health Research and Application Center, Gazi Hospital

# 2. Consent to Participate

I have read and fully understood the information provided above, including the **purpose** and scope of the study and my responsibilities as a volunteer. The study was explained to me in writing and verbally by the researcher named below, and I had the opportunity to ask questions and discuss any concerns. I received satisfactory answers, including explanations of potential risks and benefits.

I understand that I can **withdraw from the study at any time** without giving a reason, and that withdrawing will not result in any negative consequences.

Under these conditions, I voluntarily agree to participate in this study **without any pressure or coercion**.

| Participant (In own handwriting): Name-Surname: |
|---|
| Signature: |
| For Minors or Individuals Under Guardianship: Guardian Name-Surname (In own handwriting): |
| Researcher: Name-Surname: |

| Signature: | | |
|------------|-----------|------|
| | <br>••••• | <br> |